CLINICAL TRIAL: NCT05929183
Title: Efficacy and Safety Study of Neuronavigation Occipital rTMS to Improve Depressive Episodes of Bipolar Disorder in Adolescent
Brief Title: Neuronavigation rTMS to Improve Depressive Episodes of Bipolar Disorder in Adolescent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, Head of Department of Psychaitry , First Affiliated Hospital of Zhejiang University, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT20220081C-R1
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2023-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repetitive Transcranial magnetic stimulation (Active Comparator)
  Interventions: Device: Repetitive Transcranial magnetic stimulation
- Sham Repetitive Transcranial magnetic stimulation (Sham Comparator)
  Interventions: Device: Sham Repetitive Transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive Transcranial magnetic stimulation — Setting up a new target for rTMS. In the past research, the common target of rTMS in the treatment of depressive symptom was dorsolateral prefrontal cortex (DLPFC). In this study, we use high frequency rTMS in the occipital lobe are precisely targeted by navigation, by stimulating the primary visual cortex（V1), can affect the orbitofrontal cortex (OFC), which is functionally connected to V1, and thus affect the entire nerve ring pathway excitability, thereby rapidly, effectively and safely improving mood symptoms in the acute phase of bipolar depressive episode.
  After the target was determined by fMRI navigation and positioning, the subjects were subjected to rTMS for 20 minutes per day with the stimulation intensity of 10Hz and 100% of the motion threshold(MT),stimulation time of each sequence was 5 seconds, stimulation interval was 15 seconds, 3000 pulses per day for 15 days, and the total number of pulses was 45000.
  Arms: Repetitive Transcranial magnetic stimulation
Device: Sham Repetitive Transcranial magnetic stimulation — The stimulus intensity was 20% of MT in the Sham Comparator arm, and the remaining parameters were the same as the Active Comparator arm.
  Arms: Sham Repetitive Transcranial magnetic stimulation

SUMMARY:
The purpose of this study is to explore a new stimulation target and protocol for the treatment of depressive episode in adolescents with bipolar disorder through the repetitive transcranial magnetic stimulation(rTMS) under neuronavigation, and verify whether there is abnormal functional connectivity between the emotion-related brain area orbital frontal lobe (OFC) and the primary visual cortex(V1) during the depressive episode, which will contribute to further understand the relevant neural pathway and mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-28 years old, regardless of gender;
2. Meet DSM-V diagnostic criteria for bipolar depressive episodes;
3. Young Mania Rating Scale (YMRS) ≤ 6 points;
4. MARDS:12-30 points.
5. Han nationality, right-handed;
6. More than 9 years of education.

Exclusion Criteria:

1. History of severe somatic or brain organic diseases and craniocerebral trauma;
2. Abnormal brain structure or any MRI contraindications were found by magnetic resonance examination;
3. Those who do not cooperate or cannot effectively complete the experiment;
4. Drug, alcohol or other psychoactive substance abusers;
5. Pregnant, lactating or planned pregnancy.
6. Severe suicidal ideation and behavior
7. ECT or rTMS treatment was performed within six months

Ages: 14 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale（MADRS） | 0-8 weeks
  Montgomery-Asberg Depression Rating Scale (MADRS) is used to reflect the effect of antidepressant treatment and monitor the change of patients' condition. The scale is a separate scale, and the score should be based on clinical interviews. The symptoms should be asked from broad to detailed, so as to accurately score the severity. The rater must determine whether the score is on the defined score values (0,2,4,6) or between these scores (1,3,5), according to clinical practice. The scale can be used to score at any time interval.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China